CLINICAL TRIAL: NCT02643862
Title: Randomized, Controlled, Blinded, Pilot Study Using Xolair in Rush Multi Oral Immunotherapy in Multi Food Allergic Patients
Brief Title: Study Using Xolair in Rush Multi Oral Immunotherapy in Multi Food Allergic Patients
Acronym: MAP-X
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Kari Christine Nadeau, Protocol Director, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 123; U19AI104209 (NIH)
Record Dates: First submitted 2015-11-24; First posted 2015-12-31 (Estimated); Results first posted 2017-10-25 (Actual); Last update posted 2018-01-12 (Actual); Status verified 2017-12

CONDITIONS: Food Allergy
MeSH Terms: conditions — Food Hypersensitivity | interventions — Omalizumab

STUDY DESIGN:
Intervention Model Description: In a 3:1 ratio, 36* participants will receive Xolair for 16 weeks while 12* will receive corresponding placebo instead of Xolair. 12 controls will be enrolled who will receive no OIT and no Xolair. These 12 controls are not part of the randomization. The total number of participants randomized to the two arms is 48*.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- xolair (Active Comparator): Pts will be randomized to receive xolair at a 3 active:1 placebo ratio
  Interventions: Drug: Xolair
- Placebo (Placebo Comparator): This is a placebo that looks similar to Xolair and is given as a subcutaneous shot, just like Xolair
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Xolair — Xolair is a monoclonal antibody approved by the FDA for asthma and chronic urticaria
  Other Names: omalizumab
  Arms: xolair
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a pilot randomized, double-blind, placebo controlled study which will be conducted at a single center. All participants will receive oral immunotherapy for their specific food allergies (limited to 5 of those food allergens in IND 14831). In a 3:1 ratio, 36* participants will receive Xolair for 16 weeks while 12* will receive corresponding placebo instead of Xolair. 12 controls will be enrolled who will receive no OIT and no Xolair. These 12 controls are not part of the randomization. The total number of participants randomized to the two arms is 48*.

DETAILED DESCRIPTION:
We will enroll multi food allergic participants (4-55 years of age) with proven "multi food allergies". We anticipate enrolling 60 participants with allergies to, at least two foods. Participants must have food specific IgE>4kU/L for each allergen or a skin test reactivity to each food allergen ≥ 6 mm wheal diameter. We have chosen criteria associated with a very low likelihood of natural loss of food allergy for the duration of this protocol. These values of specific IgE and SPT were chosen based on the opinions of 4 experts. Participants also must have a total IgE <1500kU/L, a clinical reaction during a double blind placebo controlled food challenge (DBPCFC) with food proteins/powders to establish sensitivity to given food proteins/powders (milk, egg, peanut, almond, wheat, cashew, sesame seed, soy, walnut, hazelnut) and no clinical reaction during placebo (oat) as per CMC section of IND.

Participants will undergo a rush desensitization day at week 8 to a maximum dose of 1,250 mg total protein. Participants will be ingesting either 2 to 5 food allergens, depending on their allergy screening. They will consume home doses for two weeks based on the these results and document reactions. Upon returning to the CFRU (Clinical Food Research Unit) two weeks later, a dose escalation will be attempted. This cycle will continue until the participant reaches a maximum dose of 2,000 mg protein daily of each food allergen (two to five food allergens to be ingested by the participant). No more than 5 allergens will be given.

ELIGIBILITY:
Inclusion Criteria:

* Participant and/or parent guardian must be able to understand and provide informed consent and/or assent as applicable.
* Age 4 to 55 years with moderate to severe allergy to milk and/or egg and/or peanut and/or almond and/or wheat and/or cashew and/or sesame seed and/or soy and/or pecan and/or walnut and/or hazelnut
* ositive skin prick test result greater than or equal to 6 mm wheal diameter to each allergen OR
* ImmunoCAP IgE level >4kU/L for each allergen and
* A clinical reaction during a DBPCFC to small doses of food defined as < dose of 500 mg food protein
* No clinical reaction observed during the placebo (oat) challenge and
* If female, must have a negative urine pregnancy test on the same day (using a CLIA approved urine test)
* If female, of child-bearing potential, must agree to be compliant with a medically-approved method of contraception (please see Pregnancy section under Patient Disposition in this protocol)
* Plan to remain in the study area of the research center during the trial
* Be trained on the proper use of the Epinephrine autoinjector
* Avoid open or blinded food challenges to other allergens outside this study

Exclusion Criteria:

* Inability or unwillingness of a participant/parent/guardian to give written informed consent or comply with study protocol
* History of cardiovascular disease
* History of other chronic disease (other than asthma, atopic dermatitis, or rhinitis) requiring therapy (e.g., heart disease, diabetes) that, in the opinion of the Principal Investigator, would represent a risk to the participant's health or safety in this study or the participant's ability to comply with the study protocol
* A total IgE at screening of >1,500 kU/L
* Previous adverse reaction to Xolair
* A history of severe anaphylaxis (defined as requiring intubation or admission to an ICU) to food allergens that will be used in this study
* Unstable angina, significant arrhythmia, uncontrolled hypertension, current smokers, chronic sinusitis, or other chronic or immunological diseases that, in the judgment of the investigator, might interfere with the evaluation or administration of the test drug or pose additional risk to the participant.
* Current use of oral, intramuscular, or intravenous corticosteroids, tricyclic antidepressants, or beta-blockers (oral or topical)
* Routine use of medication that could induce adverse gastrointestinal reactions during the study
* Refusing to sign the Epinephrine autoinjector Training Form
* Pregnant or breast feeding women
* A history of oat allergy (since oat is the placebo agent in the DBPCFC), or an objective reaction to the screening DBPCFC to oat
* Unwilling to avoid all food allergen-containing items except those given as part of the OIT as well as any other food allergens you are allergic to that are not included in the 10 foods listed in the study
* Concurrent/prior use of immunomodulatory therapy (within 1 month) ie, omalizumab, non-traditional forms of allergen immunotherapy (e.g., oral or sublingual)
* Severe asthma (2007 NHLBI Criteria Steps 5 or 6) at time of enrollment
* Mild or moderate asthma (2007 NHLBI Criteria Steps 1-4) at time of enrollment with any of the following criteria met:

  * FEV1 < 80% of predicted, or FEV1/FVC < 75%, with or without controller medications (only for age 6 or greater and able to do spirometry) or
  * ICS dosing of > 220 mcg daily fluticasone (or equivalent inhaled corticosteroids based on NHLBI dosing chart) or
  * 1 hospitalization in the past year for asthma or
  * ER visit for asthma within the past six months
* Use of steroid medications (IV, IM or oral) in the following manners

  * history of daily oral steroid dosing for >1 month during the past year or
  * steroid burst course ( 5 or more days) of 1 mg/kg prednisone) course in the past 3 months or
  * >2 steroid burst courses in the past year
* Use of complementary and alternative medicine (CAM) treatment modalities (e.g., herbal remedies) for atopic and/or non-atopic disease within 90 days preceding rush desensitization at week 8or at any time .
* Inability to discontinue antihistamines for the initial day of escalation, skin testing or OFCs
* Use of investigational drugs within 24 weeks of participation
* Past or current medical problems or findings from physical assessment or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study.

Ages: 4 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Actual)
Dates: Start 2015-03-18 (Actual); Primary Completion 2016-08-20 (Actual); Study Completion 2016-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kari Nadeau, MD PhD, Study Director — Stanford University
Locations (1):
- Sean N Parker Allergy Reseach Center at Stanford University, Mountain View, California, United States

REFERENCES:
- [Derived] Manohar M, Dunham D, Gupta S, Yan Z, Zhang W, Minnicozzi S, Kirkey M, Bunning B, Roy Chowdhury R, Galli SJ, Boyd SD, Kost LE, Chinthrajah RS, Desai M, Oettgen HC, Maecker HT, Yu W, DeKruyff RH, Andorf S, Nadeau KC. Immune changes beyond Th2 pathways during rapid multifood immunotherapy enabled with omalizumab. Allergy. 2021 Sep;76(9):2809-2826. doi: 10.1111/all.14833. Epub 2021 May 29. PMID 33782956
- [Derived] Andorf S, Purington N, Block WM, Long AJ, Tupa D, Brittain E, Rudman Spergel A, Desai M, Galli SJ, Nadeau KC, Chinthrajah RS. Anti-IgE treatment with oral immunotherapy in multifood allergic participants: a double-blind, randomised, controlled trial. Lancet Gastroenterol Hepatol. 2018 Feb;3(2):85-94. doi: 10.1016/S2468-1253(17)30392-8. Epub 2017 Dec 12. PMID 29242014

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: This is a placebo that looks similar to Xolair and is given as a subcutaneous shot, just like Xolair
  Xolair: Xolair is a monoclonal antibody approved by the FDA for asthma and chronic urticaria
Period: Overall Study
Arm/Group | Xolair | Placebo
Started | 36 | 12
Completed | 36 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Xolair | Placebo | Total
Number analyzed (Participants) | 36 | 12 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 36 | 12 | 48
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 8 [5 to 11] | 7 [5 to 9] | 8 [5 to 11]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 6 | 24
  Male | 18 | 6 | 24
Region of Enrollment [Number; unit: participants]
  United States | 36 | 12 | 48

OUTCOME MEASURES:

1. Primary Outcome: Desensitization Measured by Proportion of Food Allergic (FA) Participants Who Pass a DBPCFC to 2,000 mg Protein for Each of 2 Allergens at Week 36
Description: Proportion of food allergic (FA) participants who pass a DBPCFC to 2,000 mg protein for each of 2 allergens at week 36.
  Xolair arm: 30/36 (83.3%) Placebo arm: 4/12 (33.3%)
Time Frame: 36 weeks
Population: this is an ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Xolair | Placebo
Number analyzed (Participants) | 36 | 12
Participants | 30 | 4

2. Secondary Outcome: Desensitization Measured to Increased Doses Measured by Proportion of FA Participants Who Pass a DBPCFC to 4,000 mg Each of 2 Allergens at Week 36
Description: Proportion of FA participants who pass a DBPCFC to 4,000 mg each of 2 allergens at week 36.
  Greater than 3 foods at 36 weeks for
  Xolair: 21/26 (80.8%) Placebo: 2/7 (28.6%)
Time Frame: 36 weeks
Population: We analyzed an ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Xolair | Placebo
Number analyzed (Participants) | 26 | 7
Participants | 21 | 2

ADVERSE EVENTS:
Time Frame: AEs were collected over the entire course of the active study
Description: The same definitions of AE and SAE were used as per clinicaltrials.gov
Arm/Group | Xolair | Placebo
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/12
Other Adverse Events (participants affected / at risk) | 33/36 | 12/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Xolair (N=36) | Placebo (N=12)
urticaria (Skin and subcutaneous tissue disorders) | 33 (106) | 12 (28)

LIMITATIONS AND CAVEATS:
The mechanistic 12 controls are not part of the randomization. The arms that are randomized are 48*. Mechanistic controls did not undergo therapy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes